CLINICAL TRIAL: NCT00095576
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Phase II Proof-of-Concept Study to Evaluate the Safety and Efficacy of a 3-Dose Regimen of the Merck Adenovirus Serotype 5 HIV-1 Gag/Pol/Nef Vaccine (MRK AD5 HIV-1 Gag/Pol/Nef) in Adults at High Risk of HIV-1 Infection
Brief Title: Investigation of V520 in an HIV Vaccine Proof-of-Concept Study (V520-023)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: HIV Vaccine Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V520-023; 2004_091; NCT00770549 (obsolete NCT alias)
Record Dates: First submitted 2004-11-05; First posted 2004-11-08 (Estimated); Results first posted 2011-08-15 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: AIDS; HIV Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trivalent MRKAd5 HIV-1 gag/pol/nef (Experimental): Participants randomized to receive three 1.0-ml intramuscular (IM) injections of Merck Trivalent Adenovirus Serotype 5 HIV-1 gag/pol/nef (MRKAd5 HIV-1 gag/pol/nef) Vaccine at a dose of 1.5x10^10 adenovirus genomes (Ad vg) per dose at Day 1, Week 4, and Week 26.
  Interventions: Biological: Trivalent MRKAd5 HIV-1 gag/pol/nef (1.5x10^10 ad-vg/dose)
- Placebo (Placebo Comparator): Participants randomized to receive three 1.0-ml intramuscular (IM) injections of placebo to MRKAd5 HIV-1 gag/pol/nef at Day 1, Week 4, and Week 26.
  Interventions: Drug: Comparator: placebo

INTERVENTIONS:
Biological: Trivalent MRKAd5 HIV-1 gag/pol/nef (1.5x10^10 ad-vg/dose) — Trivalent MRKAd5 HIV-1 gag/pol/nef (1.5x10^10 adenovirus genomes [ad-vg]/dose).
  This dose is equivalent to 3x10^10 vp/dose used in study V520-016.
  Other Names: V520
  Arms: Trivalent MRKAd5 HIV-1 gag/pol/nef
Drug: Comparator: placebo — Placebo to Trivalent MRKAd5 HIV-1 gag/pol/nef in three 1 mL doses at Day 1, Week 4, and Week 26 administered intramuscularly.
  Arms: Placebo

SUMMARY:
This study will test the safety and efficacy of an investigational Human Immunodeficiency Virus (HIV) vaccine. Efficacy will be measured by either prevention of HIV infection or control of HIV viral load in subjects who become HIV infected.

On September 18, 2007 the Protocol V520-023 DSMB (Data & Safety Monitoring Board) reviewed data from a planned interim analysis. These data demonstrated that the investigational vaccine candidate was not effective, and all vaccinations in the study were halted.

Participants were encouraged to continue to come to the clinic for scheduled visits and ongoing risk reduction counseling since the vaccine was not effective.

DETAILED DESCRIPTION:
No further treatment was given in V520-023, however participants were followed. V520-023 protocol ended earlier than originally planned per protocol and participants (HIV infected and uninfected) had the option of participating in an observational long term follow up protocol called V520-030/HVTN 504, which served as an extension of V520-023 and would continue through the end of 2009.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, HIV seronegative adults at high risk of acquiring HIV infection
* Cannot have previously received an investigational vaccine

Exclusion Criteria:

* In a monogamous relationship with an HIV-1 seronegative partner for > 1 year
* History of anaphylaxis and/or allergy to vaccine components, including Tris buffer, MgCl2, and polysorbate 80 (TWEEN)
* Received an immune globulin or blood derived products 3 months before injection with the first dose of vaccine/placebo or scheduled within 14 days after injection
* Previously vaccinated with a live virus vaccine within 30 days before injection with the first dose of vaccine or scheduled within 14 days after injection
* Previously vaccinated with an inactivated vaccine within 5 days before injection with the first dose of vaccine or scheduled within 14 days after injection
* Known history of immunodeficiency
* History of malignancy (with some exceptions)
* Contraindication to intramuscular (IM) injection such as anticoagulant therapy or thrombocytopenia
* Female subject who is pregnant or breast feeding, or expecting to conceive or donate eggs through Week 30 of the study
* Male subject who is planning to impregnate or provide sperm donation through Week 30 of the study
* Previously received an investigational HIV vaccine
* Has active drug or alcohol abuse or dependence that would interfere with adherence to study requirements, or endanger the subject's health while on the study
* Has a condition that might endanger the subject's health or interfere with the evaluation of the study objectives

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3000 (Actual)
Dates: Start 2004-11; Primary Completion 2007-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Buchbinder SP, Mehrotra DV, Duerr A, Fitzgerald DW, Mogg R, Li D, Gilbert PB, Lama JR, Marmor M, Del Rio C, McElrath MJ, Casimiro DR, Gottesdiener KM, Chodakewitz JA, Corey L, Robertson MN; Step Study Protocol Team. Efficacy assessment of a cell-mediated immunity HIV-1 vaccine (the Step Study): a double-blind, randomised, placebo-controlled, test-of-concept trial. Lancet. 2008 Nov 29;372(9653):1881-1893. doi: 10.1016/S0140-6736(08)61591-3. Epub 2008 Nov 13. PMID 19012954
- [Derived] Janes H, Friedrich DP, Krambrink A, Smith RJ, Kallas EG, Horton H, Casimiro DR, Carrington M, Geraghty DE, Gilbert PB, McElrath MJ, Frahm N. Vaccine-induced gag-specific T cells are associated with reduced viremia after HIV-1 infection. J Infect Dis. 2013 Oct 15;208(8):1231-9. doi: 10.1093/infdis/jit322. Epub 2013 Jul 21. PMID 23878319
- [Derived] Duerr A, Huang Y, Buchbinder S, Coombs RW, Sanchez J, del Rio C, Casapia M, Santiago S, Gilbert P, Corey L, Robertson MN; Step/HVTN 504 Study Team. Extended follow-up confirms early vaccine-enhanced risk of HIV acquisition and demonstrates waning effect over time among participants in a randomized trial of recombinant adenovirus HIV vaccine (Step Study). J Infect Dis. 2012 Jul 15;206(2):258-66. doi: 10.1093/infdis/jis342. Epub 2012 May 4. PMID 22561365
- [Derived] Barnabas RV, Wasserheit JN, Huang Y, Janes H, Morrow R, Fuchs J, Mark KE, Casapia M, Mehrotra DV, Buchbinder SP, Corey L; NIAID HIV Vaccine Trials Network. Impact of herpes simplex virus type 2 on HIV-1 acquisition and progression in an HIV vaccine trial (the Step study). J Acquir Immune Defic Syndr. 2011 Jul 1;57(3):238-44. doi: 10.1097/QAI.0b013e31821acb5. PMID 21860356
- [Derived] Fitzgerald DW, Janes H, Robertson M, Coombs R, Frank I, Gilbert P, Loufty M, Mehrotra D, Duerr A; Step Study Protocol Team. An Ad5-vectored HIV-1 vaccine elicits cell-mediated immunity but does not affect disease progression in HIV-1-infected male subjects: results from a randomized placebo-controlled trial (the Step study). J Infect Dis. 2011 Mar 15;203(6):765-72. doi: 10.1093/infdis/jiq114. PMID 21343146

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3000 participants were enrolled and randomized in the study. However, only 2979 received study vaccination, and are included in the started population.
  V520-023 was terminated early based on findings at a planned interim analysis and subjects were encouraged to participate in the V520-030 rollover study for additional long term follow up.
Period: Overall Study
Arm/Group | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef | Placebo
Started | 1484 | 1495
VACCINATED AT VISIT 2 (Dose 1) | 1484 | 1495
VACCINATED AT VISIT 4 (Dose 2) | 1426 | 1443
VACCINATED AT VISIT 7 (Dose 3) | 1328 | 1361
Completed | 9 (Subjects not completing entire study were eligible for observational long term follow up in V520-030) | 14 (Subjects not completing entire study were eligible for observational long term follow up in V520-030)
Not Completed | 1475 | 1481
Not completed — Adverse Event | 5 | 3
Not completed — Lost to Follow-up | 233 | 229
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 34 | 47
Not completed — Option to switch to a rollover study | 1097 | 1099
Not completed — Site terminated | 75 | 67
Not completed — Subject moved | 30 | 36

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef | Placebo | Total
Number analyzed (Participants) | 1484 | 1495 | 2979
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (7.8) [18 to 46] | 30.2 (8.13) [18 to 45] | 30.1 (7.97) [18 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 565 | 570 | 1135
  Male | 919 | 925 | 1844

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Adverse Experiences
Description: Number of participants with non-serious AEs with an incidence cut-off of 5% (>5% in at least one treatment group) and number of participants with >1 SAE following administration of study vaccine.
  AEs collected include serious and non-serious systemic AEs, and injection-site AEs. All systemic AEs were collected up to 14 days after any vaccine dose, and serious AEs were collected for the entire study period (up to Week 210).
  Injection-site AEs are any swelling, redness, pain or tenderness at the injection site. All injection site AEs were collected up to Day 4 after any vaccine dose.
Time Frame: Day 1 to End of Study (Week 210 for HIV uninfected participants and Week 338 for HIV infected participants)
Measure: Number; unit: Participants
Arm/Group | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef | Placebo
Number analyzed (Participants) | 1484 | 1495
Participants
  With non-serious adverse events (NSAE) | 1221 | 946
  With no non-serious adverse events | 263 | 549
  With serious adverse events | 19 | 17
  With no serious adverse events | 1465 | 1478

2. Primary Outcome: Number of Participants With Laboratory Adverse Experiences
Description: Number of participants with laboratory adverse experiences with an incidence cut-off of 5% (events occurring > 5% in at least one treatment group) following administration of the first dose of study vaccine.
  Laboratory AEs were based on a grading system considering the severity of abnormal laboratory values in participants and reflect any unfavorable and unintentional change in function, or chemistry of the body.
  All laboratory AEs were collected up to 14 days after any vaccine dose.
Time Frame: Day 1 to Week 208
Measure: Number; unit: Participants
Arm/Group | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef | Placebo
Number analyzed (Participants) | 1484 | 1495
Participants | 0 | 0

3. Primary Outcome: Number of Participants With HIV-1 Infections
Description: The number of participants with HIV-1 infections was to be determined with a periodic HIV-1 screening test to detect antibodies to recombinant HIV-1 envelope protein in the participants' serum.
Time Frame: Day 1 to End of Study (Week 210 for HIV uninfected participants and Week 338 for HIV infected participants)
Population: An interim analysis for this study showed that the MRK Ad5 HIV-1 gag/pol/nef vaccine used in this study was not efficacious; therefore, this outcome measure was not analyzed and only a high level summary of the safety data was performed.
Arm/Group | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef | Placebo
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: HIV-1 Viral Load in Infected Participants
Description: Plasma HIV-1 viral RNA was to be measured using a ribonucleic acid polymerase chain reaction (RNA PCR) on the last archived sample, and at Weeks 1, 2, 8, 12, and 26 post-HIV-1 infection, and subsequently every 6 months.
Time Frame: Day 1 to End of Study (Week 210 for HIV uninfected participants and Week 338 for HIV infected participants)
Population: as for outcome 3
Arm/Group | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef | Placebo
Serious Adverse Events (participants affected / at risk) | 19/1484 | 17/1495
Other Adverse Events (participants affected / at risk) | 1221/1484 | 946/1495
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef (N=1484) | Placebo (N=1495)
Anemia aggravated (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Congenital cardiovascular anomaly (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
Hypoplastic left heart syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Unspecified congenital anomaly of heart (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Acute diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Rigors (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Shunt infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 1 (1) | 0 (0)
Vulval abscess (Infections and infestations) | 1 (1) | 0 (0)
Asbestosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Slipped disc (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine fibroids (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Depression aggravated (Psychiatric disorders) | 0 (0) | 1 (1)
Depressive episode (Psychiatric disorders) | 1 (1) | 0 (0)
Manic episode (Psychiatric disorders) | 0 (0) | 1 (1)
Polysubstance dependence (Psychiatric disorders) | 1 (1) | 0 (0)
Substance abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Kidney stone (Renal and urinary disorders) | 1 (1) | 0 (0)
Exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef (N=1484) | Placebo (N=1495)
Diarrhoea (Gastrointestinal disorders) | 156 (195) | 148 (182)
Nausea (Gastrointestinal disorders) | 94 (114) | 75 (87)
Fatigue (General disorders) | 170 (218) | 120 (149)
Fever (General disorders) | 376 (631) | 309 (548)
General body pain (General disorders) | 76 (98) | 23 (26)
Injection site erythema (General disorders) | 317 (448) | 143 (197)
Injection site pain (General disorders) | 961 (1862) | 475 (702)
Injection site swelling (General disorders) | 337 (511) | 115 (149)
Injection site tenderness (General disorders) | 271 (374) | 81 (92)
Headache (Nervous system disorders) | 461 (734) | 394 (631)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 83 (96) | 83 (90)

LIMITATIONS AND CAVEATS:
The DSMB (Data & Safety Monitoring Board) reviewed interim data which demonstrated that the investigational vaccine was not effective, and all vaccinations were halted. Long term follow up was available for participants in V520-030.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
As this study is part of a multicenter trial, publications derived from this study should include input from the principal investigator, his/her colleagues, the other investigators in this trial, and SPONSOR personnel.

The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. SPONSOR review can be expedited to meet publication guidelines.